CLINICAL TRIAL: NCT03116932
Title: Evaluating the Feasibility and Acceptability of Implementing a PrEP Program in PR-CoNCRA (San Juan, Puerto Rico)- Part A
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Puerto Rico Community Network for Clinical Research on AIDS (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Vivian Tamayo-Agrait, MD, Principal Investigator, Puerto Rico Community Network for Clinical Research on AIDS
Other Study IDs: Puerto Rico PrEP Study-Part A
Record Dates: First submitted 2017-03-27; First posted 2017-04-17 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: HIV/AIDS
Keywords: HIV prevention, high risk MSM, PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Dried Blood Spots are obtained at 2 time points for participants in part B in order to assess adequate drug levels are retained for bulk shipping for processing at collaborating lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Part A - high risk MSM: Part A will consist of a descriptive analysis of the acceptability and knowledge on the topic of PrEP of the individuals that undergo routine HIV testing and counseling in study facilities or through outreach activities.
  Part A will be focused only on high risk MSM. For this part of the study, 225 high risk will be interviewed to understand the knowledge and acceptability of PrEP in this population in Puerto Rico.
  Interventions: Behavioral: PrEP knowledge and acceptability questionnaire

INTERVENTIONS:
Behavioral: PrEP knowledge and acceptability questionnaire — This questionnaire consists of 187 items and evaluates socio-demographic variables, sex conducts, PrEP knowledge and PrEP acceptability.

SUMMARY:
The target population for this project will be men-who-have-sex-with-men (MSM) at high risk of HIV acquisition

DETAILED DESCRIPTION:
225 high risk MSM will be interviewed to understand the knowledge and acceptability of pre-exposure prophylaxis (PrEP) in this population in Puerto Rico. A 187 item questionnaire will administered which will evaluate socio-demographic information, sexual conducts, PrEP knowledge and PrEP acceptability.

ELIGIBILITY:
INCLUSION CRITERIA;

Study subjects who meet the following inclusion criteria will be considered for enrollment for Part A:

1. age 21 years or older
2. understand and sign the informed consent form and willing to participate in the study
3. male or transgender female
4. has one of the following risk factors:

   * a high risk MSM as defined by:
   * having unprotected sexual intercourse with at least two male partners in the past 6 months, or
   * diagnosed with an STI in the past 6 months.

PART A - EXCLUSION CRITERIA:

Subjects with any of the following will not be considered for enrollment in Part A:

1. Age younger than 21 years old
2. Unable or unwilling to provide an informed consent
3. Female gender at birth
4. Do not meet the high risk criteria

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male-to-female transgender subjects are eligible for enrollment
Study Population: 225 high risk men who have sex with men, HIV- subjects, 21 years or older , will be enrolled in Part A
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
PrEP acceptability using a PrEP knowledge and acceptability questionnaire. | One visit
  Measure the degree of acceptance of PrEP in the study subjects
PrEP knowledge using a PrEP knowledge and acceptability questionnaire. | One visit
  Measure the level of education of the study subjects in the topic of PrEP using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Tamayo-Agrait, MD, Principal Investigator — 787-753-9443
Locations (1):
- Puerto Rico Community Network for Clinical Research on AIDS (PR-CoNCRA), San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided